CLINICAL TRIAL: NCT06404931
Title: Transvaginal Human Acellular Dermal Matrix and Sacrospinous Fixation for Anterior and Apical Prolapse Treatment in Patients With Hiatal Ballooning or Levator Ani Injury: a Randomized Pilot Trial
Brief Title: Transvaginal Human Acellular Dermal Matrix for Prolapse Treatment
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Mutua de Terrassa (Other)
Collaborators: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other); Germans Trias i Pujol Hospital (Other); Hospital Arnau de Vilanova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Mesh in prolapse treatment
Record Dates: First submitted 2024-03-08; First posted 2024-05-08 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2025-01

CONDITIONS: Prolapse; Female; Prolapse Genital; Prolapse Uterovaginal
MeSH Terms: conditions — Prolapse | interventions — Hysterectomy, Vaginal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Vaginal hysterectomy plus anterior colporrhaphy (Sham Comparator): Vaginal hysterectomy plus anterior colporrhaphy
  Interventions: Procedure: Vaginal hysterectomy plus anterior colporrhaphy
- Vaginal hysterectomy plus sacrospinous fixation with Anchorsure® device (Sham Comparator): Vaginal hysterectomy plus sacrospinous fixation with Anchorsure® device
  Interventions: Procedure: Vaginal hysterectomy plus sacrospinous fixation with Anchorsure® device
- Vaginal hysterectomy plus matrix reinforcement and sacrospinous fixation with Anchorsure® device (Experimental): Vaginal hysterectomy plus matrix reinforcement and sacrospinous fixation with Anchorsure® device
  Interventions: Procedure: Vaginal hysterectomy plus matrix reinforcement and sacrospinous fixation with Anchorsure® device

INTERVENTIONS:
Procedure: Vaginal hysterectomy plus matrix reinforcement and sacrospinous fixation with Anchorsure® device — Vaginal hysterectomy plus matrix reinforcement and sacrospinous fixation with Anchorsure® device
  Arms: Vaginal hysterectomy plus matrix reinforcement and sacrospinous fixation with Anchorsure® device
Procedure: Vaginal hysterectomy plus anterior colporrhaphy — Vaginal hysterectomy plus anterior colporrhaphy
  Arms: Vaginal hysterectomy plus anterior colporrhaphy
Procedure: Vaginal hysterectomy plus sacrospinous fixation with Anchorsure® device — Vaginal hysterectomy plus sacrospinous fixation with Anchorsure® device
  Arms: Vaginal hysterectomy plus sacrospinous fixation with Anchorsure® device

SUMMARY:
This is a randomised study in which we compare the effectiveness of three different procedures in mending symptomatic anterior and apical prolapse in patients who are candidates to receive surgery.

They will be randomly assigned in a ratio 1:1:1 to three different groups who will have assigned three different kinds of surgery. In the patients of the first group a classic vaginal hysterectomy with anterior colporrhaphy will be practised. Patients who belong to group two will undergo a vaginal hysterectomy followed by placement of an acellular dermal matrix from cadaveric donors (hADM) for anterior reinforcement and sacrospinous fixation with Anchorsure® device (Neomedic trade mark (TM) International, Spain). Finally, patients from group three will have vaginal hysterectomy followed by sacrospinous fixation with Anchorsure® alone .

Patients will be followed-up at 4 weeks, 6 months, 12 months and annually till 36 months to evaluate relapses and possible complications.

DETAILED DESCRIPTION:
Eligible patients will be women with symptomatic anterior and apical prolapse with hiatal ballooning or levator ani injury eligible for vaginal surgical treatment.

At the time of the indication for surgery, anatomical severity of the prolapse (according to the Pelvic Organ Prolapse Quantification System (POP-Q) scale) and the symptoms of prolapse and sexual function, as well as their impact on the quality of life of the patient, are evaluated using validated questionnaires "Pelvic Floor Impact Questionnaire (PFIQ)", "Pelvic organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12)"and "European Quality of Life-5 Dimensions Questionnaire (EQ5D)". Anatomical severity of the prolapse will be also evaluated by ecography described as follows.

Three-dimensional 3D/4D transperineal ultrasound (TPS) will be performed using a GE Voluson® ultrasound system (GE Medical Systems) with a RAB 8-4-MHz transducer at an acquisition angle of 85°.

TPS will be performed with the probe covered with a powder-free glove and applied in the midsagittal plane to the introitus using moderate pressure. Volumes are acquired at rest, on maximum pelvic floor muscle contractility and during maximal Valsalva maneuver. Patients perform Valsalva for at least 5 s, and the best of three volumes is used for analysis. Using visual biofeedback, an attempt is made to correct for levator co-activation by requesting the women observe the narrowing and widening of the levator hiatus during the maneuvers.

3D volumes are measured offline using GE 4 Dimension View (GE Medical Systems). Using the best Valsalva maneuver, pelvic organ descent measurements are obtained relative to a horizontal line from the inferior margin of the pubic symphysis. Levator hiatal area is assessed in the plane of minimal hiatal dimensions.

Surgical indication will be determined by gynaecologists and the decision will be clearly dissociated from the decision of study inclusion. Therefore, the performance of the study should not modify the habits of surgical indication by the doctors.

The study will be a single-blinded study, as it is impossible to blind the health care workers involved for the surgical procedure to which the woman is randomized. The physician evaluating the patients during the follow-up will be blinded about the group the patients were randomized to.

Women will be randomly assigned after consenting for participation in the study, by means of an interactive response technology system in a 1:1:1 ratio to receive surgical treatment with vaginal hysterectomy followed by hADM anterior reinforcement and sacrospinous fixation with Anchorsure® device (NeomedicTM International, Spain), vaginal hysterectomy followed by sacrospinous fixation with Anchorsure® alone or classic vaginal hysterectomy with anterior colporrhaphy. A sacrospinous fixation-alone group was included to assess the impact of this technique in the principal surgery group. Patients will be followed-up at 4 weeks, 6 months, 12 months and annually till 36 months.

Anatomical results will be evaluated by a member of the team blinded to the surgery performed during follow-up visits after surgery and by 3D ultrasound of the pelvic floor. Functional results are evaluated using the validated questionnaires performed prior to surgery done by the patients during follow-up visits after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Women with symptomatic POP with indication of vaginal surgery.
* Women with hiatal ballooning or levator ani injury evaluated by 3D pelvic floor ultrasound.
* Women ≥18 years old.
* Women wishing to complete a 36-month follow-up.
* Understand and accept the study procedures and sign the informed consent.

Exclusion Criteria:

* Women with previous pelvic floor or prolapse surgery
* Women with POP grade IV
* Women with chronic pelvic pain.
* Not being able to understand the nature of the study and/or the procedures to be followed.
* Not signing the informed consent

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence of anatomical anterior vaginal wall prolapse | 36 months
  Defined as point Ba POP-Q stage ≥II by clinical examination

SECONDARY OUTCOMES:
Difference between groups in anatomical prolapse | 36 moths
  Defined as point C POP-Q stage ≥II by clinical examination
Differences between groups in symptomatic recurrence | 36 months
  Evaluated by Pelvic Floor Impact Questionnaire. Minimum value: 0. Maximum value: 300. The higher the value worse is the outcome
Differences between groups in quality of Life | 36 months
  Evaluated by European Quality of Life-5 Dimensions Questionnaire. Minimum value: 0. Maximum value: 1. The higher the value the worse is the outcome
Differences between groups in sexual functioning. | 36 months
  Evaluated by Pelvic organ Prolapse/Urinary Incontinence Sexual Questionnaire. Minimum value: 0. Maximum value: 100. The higher the value the worse is the outcome
Differences between groups in hospital stay | 36 months
  Evaluated by number of days of hospital stay
Differences between groups in operative time | 36 months
  Evaluated by minutes of duration of surgery
Differences between groups in surgical complication rate. | 36 months
  Monitoring of development of hematoma, urologic lesion, need for blood transfusion, suture dehiscence, pain, infection and mesh extrusion
Differences between groups in reintervention rate | 36 months
  Reintervention will be done in cases of symptomatic recurrence of the compartment previously treated or development of another prolapse.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Mutua de Terrassa, Terrassa, Spain

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in the publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).

REFERENCES:
- [Background] Flynn BJ, Webster GD. Surgical management of the apical vaginal defect. Curr Opin Urol. 2002 Jul;12(4):353-8. doi: 10.1097/00042307-200207000-00015. PMID 12072658
- [Background] Unger CA, Barber MD. Vaginal Mesh in Pelvic Reconstructive Surgery: Controversies, Current Use, and Complications. Clin Obstet Gynecol. 2015 Dec;58(4):740-53. doi: 10.1097/GRF.0000000000000148. PMID 26512439
- [Background] NHS Improvement, NHS England. Letter to Acute Trust CEOs and Medical Directors. 2018;(July 2017). Available from: www.england.nhs.uk
- [Background] Salzberg CA. Nonexpansive immediate breast reconstruction using human acellular tissue matrix graft (AlloDerm). Ann Plast Surg. 2006 Jul;57(1):1-5. doi: 10.1097/01.sap.0000214873.13102.9f. PMID 16799299
- [Background] Guo X, Mu D, Gao F. Efficacy and safety of acellular dermal matrix in diabetic foot ulcer treatment: A systematic review and meta-analysis. Int J Surg. 2017 Apr;40:1-7. doi: 10.1016/j.ijsu.2017.02.008. Epub 2017 Feb 14. PMID 28232031
- [Background] Menon NG, Rodriguez ED, Byrnes CK, Girotto JA, Goldberg NH, Silverman RP. Revascularization of human acellular dermis in full-thickness abdominal wall reconstruction in the rabbit model. Ann Plast Surg. 2003 May;50(5):523-7. doi: 10.1097/01.SAP.0000044252.76804.6B. PMID 12792544
- [Background] Salzberg CA, Ashikari AY, Koch RM, Chabner-Thompson E. An 8-year experience of direct-to-implant immediate breast reconstruction using human acellular dermal matrix (AlloDerm). Plast Reconstr Surg. 2011 Feb;127(2):514-524. doi: 10.1097/PRS.0b013e318200a961. PMID 21285756
- [Background] Griffey S, Schwade ND, Wright CG. Particulate dermal matrix as an injectable soft tissue replacement material. J Biomed Mater Res. 2001;58(1):10-5. doi: 10.1002/1097-4636(2001)58:13.0.co;2-e. PMID 11152992
- [Background] Botros SM, Sand PK, Beaumont JL, Abramov Y, Miller JJ, Goldberg RP. Arcus-anchored acellular dermal graft compared to anterior colporrhaphy for stage II cystoceles and beyond. Int Urogynecol J Pelvic Floor Dysfunct. 2009 Oct;20(10):1265-71. doi: 10.1007/s00192-009-0933-7. Epub 2009 Jun 17. PMID 19533005
- [Background] Clemons JL, Myers DL, Aguilar VC, Arya LA. Vaginal paravaginal repair with an AlloDerm graft. Am J Obstet Gynecol. 2003 Dec;189(6):1612-8; discussion 1618-9. doi: 10.1016/s0002-9378(03)00929-3. PMID 14710083
- [Background] Ward RM, Sung VW, Clemons JL, Myers DL. Vaginal paravaginal repair with an AlloDerm graft: Long-term outcomes. Am J Obstet Gynecol. 2007 Dec;197(6):670.e1-5. doi: 10.1016/j.ajog.2007.08.067. PMID 18060976
- [Background] Chung SY, Franks M, Smith CP, Lee JY, Lu SH, Chancellor M. Technique of combined pubovaginal sling and cystocele repair using a single piece of cadaveric dermal graft. Urology. 2002 Apr;59(4):538-41. doi: 10.1016/s0090-4295(01)01611-9. PMID 11927309
- [Background] Miklos JR, Kohli N, Moore R. Levatorplasty release and reconstruction of rectovaginal septum using allogenic dermal graft. Int Urogynecol J Pelvic Floor Dysfunct. 2002;13(1):44-6. doi: 10.1007/s001920200009. PMID 11999206
- [Background] Kohli N, Miklos JR. Dermal graft-augmented rectocele repair. Int Urogynecol J Pelvic Floor Dysfunct. 2003 Jun;14(2):146-9. doi: 10.1007/s00192-002-1013-4. Epub 2003 Feb 13. PMID 12851761
- [Background] Perez ML, Castells-Sala C, Lopez-Chicon P, Nieto-Nicolau N, Aiti A, Farinas O, Casaroli-Marano RP, Porta O, Vilarrodona A. Fast protocol for the processing of split-thickness skin into decellularized human dermal matrix. Tissue Cell. 2021 Oct;72:101572. doi: 10.1016/j.tice.2021.101572. Epub 2021 Jun 4. PMID 34119882
- [Background] Pero M, Casani L, Castells-Sala C, Perez ML, Moga Naranjo E, Juan-Babot O, Alserawan De Lamo L, Lopez-Chicon P, Vilarrodona Serrat A, Badimon L, Porta Roda O. Rabbit as an animal model for the study of biological grafts in pelvic floor dysfunctions. Sci Rep. 2021 May 18;11(1):10545. doi: 10.1038/s41598-021-89698-z. PMID 34006889
- [Background] Curtiss N, Duckett J. A long-term cohort study of surgery for recurrent prolapse comparing mesh augmented anterior repairs to anterior colporrhaphy. Gynecol Surg. 2018;15(1):1. doi: 10.1186/s10397-017-1035-z. Epub 2018 Jan 10. PMID 29375283
- [Background] Altman D, Vayrynen T, Engh ME, Axelsen S, Falconer C; Nordic Transvaginal Mesh Group. Anterior colporrhaphy versus transvaginal mesh for pelvic-organ prolapse. N Engl J Med. 2011 May 12;364(19):1826-36. doi: 10.1056/NEJMoa1009521. PMID 21561348
- [Background] Wong NKL, Cheung RYK, Lee LL, Wan OYK, Choy KW, Chan SSC. Women with advanced pelvic organ prolapse and levator ani muscle avulsion would significantly benefit from mesh repair surgery. Ultrasound Obstet Gynecol. 2021 Apr;57(4):631-638. doi: 10.1002/uog.23109. PMID 32898286
- [Background] Rodrigo N, Wong V, Shek KL, Martin A, Dietz HP. The use of 3-dimensional ultrasound of the pelvic floor to predict recurrence risk after pelvic reconstructive surgery. Aust N Z J Obstet Gynaecol. 2014 Jun;54(3):206-11. doi: 10.1111/ajo.12171. Epub 2014 Feb 18. PMID 24576013
- [Background] Vollebregt A, Fischer K, Gietelink D, van der Vaart CH. Primary surgical repair of anterior vaginal prolapse: a randomised trial comparing anatomical and functional outcome between anterior colporrhaphy and trocar-guided transobturator anterior mesh. BJOG. 2011 Nov;118(12):1518-27. doi: 10.1111/j.1471-0528.2011.03082.x. Epub 2011 Aug 22. PMID 21864325
- [Background] Dietz HP. Ultrasound imaging of the pelvic floor. Part II: three-dimensional or volume imaging. Ultrasound Obstet Gynecol. 2004 Jun;23(6):615-25. doi: 10.1002/uog.1072. PMID 15170808